CLINICAL TRIAL: NCT03972592
Title: 0.1% Topical Sirolimus in the Treatment of Cutaneous Microcystic Lymphatic Malformations in Children and Adults: Phase II, Split-body Randomized, Double-blind, Vehicle-controlled Clinical Trial
Brief Title: Topical Sirolimus in Cutaneous Lymphatic Malformations
Acronym: TOPICAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRN17-AM / TOPICAL (DR180115); 2018-001359-11 (EudraCT Number)
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Vascular Malformations; Lymphatic Malformation
Keywords: Cutaneous Microcystic Lymphatic Malformations
MeSH Terms: conditions — Vascular Malformations; Lymphatic Abnormalities | interventions — Sirolimus; calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: Split-body randomised, double-blind, vehicle-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, parents, nurses and investigators will be blinded for the treatment allocated to each area of the CMLM, during the first step of the study (until week 12, where primary endpoint will be assessed). To ensure the double blinding, both areas will be randomized, and the topical treatments (sirolimus and vehicle) to be applied will have similar packaging. Their appearance is similar, thus the active drug (topical sirolimus) and vehicle cannot be distinguished at drug allocation. Furthermore, the consistency of the creams is similar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical sirolimus (Experimental): The experimental group will consist in one area of the CMLM (almost half of it) that will receive 0.1% sirolimus preparation. This product will be applied 1/day on the randomly allocated area, by a nurse at home, during 12 weeks.
  Interventions: Drug: Topical 0.1% Sirolimus
- Vehicle (Placebo Comparator): The control group will consist in the other half area of the CMLM, that will receive the same vehicle than the one used in the topical 0.1% sirolimus preparation. It will be applied 1/day in the corresponding area by a nurse, at home, during 12 weeks.
  Interventions: Drug: Topical Vehicle

INTERVENTIONS:
Drug: Topical 0.1% Sirolimus — The formulation is 0.03 g rapamycin, 1.5 g Transcutol, Quantum Satis (QS) 30g Excipial® hydrocream, corresponding to a concentration at 0.1%. The cream will be packaged in 30 ml aluminium tubes.
  Other Names: Verum
  Arms: Topical sirolimus
Drug: Topical Vehicle — The same vehicle than the one used in the topical 0.1% sirolimus preparation will be used for the other half area of CMLM, i.e. Excipial® hydrocream. It will be packaged to maintain the double blind way of this trial and will be undistinguishable from the sirolimus cream.
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
Cutaneous microcystic lymphatic malformations (CMLMs) are rare conditions of children and adults resulting from abnormal embryologic development of lymphatic vessels. They present as clusters of vesicles full of lymph and blood of various extent. They ooze and bleed, inducing maceration, esthetic impairment, scars, pain, bacterial infections and impaired quality of life. Currently, treatments for CMLMs are disappointing, and their management is challenging. Sirolimus is an inhibitor of mammalian target of rapamycin (mTOR), a serine/threonine protein kinase involved in cell growth and proliferation, cellular metabolism, autophagy and angio-lymphangiogenesis. Topical sirolimus, known to be efficient and well tolerated in cutaneous angiofibromas linked to tuberous sclerosis, has recently been reported effective in few reports of patients with CMLMs. The objective of this trial is to compare the efficacy and safety of a 12-week application of 0.1% topical sirolimus versus topical vehicle in CMLMs in children and adults.

DETAILED DESCRIPTION:
This blinded multicentre split body randomized controlled phase 2 trial aims to include 50 patients ≥ 6 years old who have a primary CMLM without an underlying malformation.

The CMLM will be divided into 2 equal areas of the same severity that will be randomly allocated to 0.1% topical sirolimus or topical vehicle for 12 weeks. During the double-blind 12-week period, both topical products will be applied by a nurse to avoid inter-group contamination and for better compliance.

At the end of the 12-week period, the patient/parent will treat the whole area of CMLM with 0.1% topical sirolimus on remaining lesions, for 8 more weeks. Patients will also be seen at week 20 (treatment will be stopped) and at month 12 to evaluate long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 6 years
* Updated immunization schedule
* Diagnosis of primary cutaneous microcystic lymphatic malformation (CMLM) confirmed by histopathological or dermoscopic examination, with or without an underlying malformation or a syndromic malformation (Protée syndrome for instance), responsible for impairment (oozing, bleeding and/or pain)
* CMLM ≥ 20 cm2, that can be divided into 2 parts of similar severity
* Informed, written consent of the subject and his/her parents if < 18 years
* Rights to French social security (including CMU)

Exclusion Criteria:

* Patients with lymphatic malformation requiring a continued background therapy (involving deep organs)
* Secondary lymphatic malformations (lymphangiectasia post-radiotherapy, etc)
* Previous treatment with oral or topical mTOR inhibitors within 12 months before inclusion
* Previous treatment with oral or topical steroids within 10 days before inclusion
* Immunosuppression (immunosuppressive disease or immunosuppressive treatment)
* Ongoing neoplasia
* Active chronic infectious disease (Hepatitis B Virus, Hepatitis C Virus, Human Immunodeficiency Virus, etc)
* Local fungal, viral (Herpes Simplex Virus, Varicella Zoster Virus, etc) or bacterial infection on the site of the CMLM (based on clinical examination)
* Skin necrosis
* Known allergy to one of the components of the topical sirolimus preparation or vehicle
* Women of child-bearing potential (including teenagers) not using a reliable contraceptive method until the end of the study
* Pregnant or breastfeeding women
* Subject already involved in another therapeutic trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a 12-week application period of 0.1% topical sirolimus in cutaneous microcystic lymphatic malformation versus topical vehicle | Week 12
  PGA (Physician Global Assessment) score assessed by the investigator physician (blinded from the treatment). PGA score ranges from 0 (clear) to 5 (severe lesions), and is commonly used in several dermatologic conditions. For each patient, PGA of the area treated with the intervention (0.1% topical sirolimus) will be compared to PGA of the area treated with topical vehicle (inactive comparator)

SECONDARY OUTCOMES:
Efficacy of 0.1% topical sirolimus in cutaneous microcystic lymphatic malformation versus topical vehicle | Day 1, Week 6, Week 20, Month 12
  PGA (Physician Global Assessment) score assessed by the investigator physician (blinded from the treatment). PGA score ranges from 0 (clear) to 5 (severe lesions), and is commonly used in several dermatologic conditions. For each patient, PGA of the area treated with the intervention (0.1% topical sirolimus) will be compared to PGA of the area treated with topical vehicle (inactive comparator)
Efficacy of 0.1% topical sirolimus vs vehicle regarding each of the following complications of the CMLM: oozing, bleeding, erythema, and thickness | Day 1, Week 12, Week 20, Month 12
  Assessment by the investigator blinded to treatment with a visual analog scale (VAS) from 0 to 10 (0: no improvement, 10: recovery)
Number of independent experts who correctly identify which area among both received the active treatment for each patient on the basis of standardised photographs | Day1, Week 12
  Standardized photographs will be performed at baseline and week 12: the experts will have to identify, at the end of the study, which area among both received the active treatment. In case of disagreement, a consensus will be reached between both experts; if consensus is not reached, a third expert will be sought for final decision. Interpretation by dermatologic experts (i.e correct identification of intervention/vehicle treated area) will be considered as correct or false, and the proportion of correct interpretation will be estimated. The proportion of correct interpretation will be compared to the theoretical 50% value, corresponding to a random assessment. Five photographs will be taken: 1) one of the patient including the malformation 2) one of the malformation (distance of 50 cm), 3) one of the malformation (distance of 15 cm), 4) profile photography and finally 5) three quarter view.
Global self-reported efficacy of topical sirolimus vs vehicle (with help of parents in case of children under 16 years) | Week 12, Week 20, Month 12
  Self-assessment of the global improvement of CMLM in both areas using a VAS (Visual Analog Scale) from 0 to 10 (0 no improvement and 10 recovery)
Functional and esthetic impairments (self-reported with help of parents in case of children under 16 years) | Day1, Week 20, Month 12
  Using a VAS (Visual Analog Scale) from 0 to 10 (0 no improvement and 10 recovery)
Pain linked to the CMLM (with help of parents in case of children under 16 years) | Day1, Week 20, Month 12
  Using a VAS (Visual Analog Scale) from 0 to 10 (0 no pain and 10 worst imaginable pain)
Effect on quality of life | Day 1, Week 20, Month 12
  Self-assessment of quality of life using the validated DLQI (Dermatology Life Quality Index) scale, or Child-DLQI for children (equal ou under 16 years old) from 0 to 30 (0 no impact on quality of life and 30 maximum impact on quality of life)
Evaluation of systemic passage of sirolimus by dosage of serum level of sirolimus | Week 6, Week 12, Week 20, +/- Week 16 (if CMLM ≥ 30*30 cm and/or ≥900 cm2)
  Dosage of serum level of sirolimus
Number of patients with biological adverse events and total number of biological adverse events (to assess the biological tolerance of topical sirolimus) | Baseline, Week 12, Week 20
  Number of patients with biological adverse events and total number of biological adverse events (blood samples at baseline, week 12 and week 20)
Number of patients with clinical adverse events and total number of clinical adverse events (to assess the clinical tolerance of topical sirolimus) | Week 6, Week 12, Week 20
  Number of patients with clinical adverse events and total number of clinical adverse events (record of local and general adverse events)

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - ANGERS, Angers
  - BORDEAUX, Bordeaux
  - LYON AD, Bron
  - LYON PED, Bron
  - CAEN, Caen
  - DIJON, Dijon
  - Marseille, Marseille
  - Montpellier, Montpellier
  - NANTES, Nantes
  - NICE, Nice
  - Lariboisiere, Paris
  - NECKER, Paris
  - QUIMPER, Quimper
  - RENNES, Rennes
  - TOULOUSE, Toulouse
  - TOURS, Tours
  - NANCY, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leducq S, Caille A, Barbarot S, Beneton N, Bessis D, Boccara O, Bursztejn AC, Chiaverini C, Dompmartin A, Droitcourt C, Gissot V, Goga D, Guibaud L, Herbreteau D, Le Touze A, Leaute-Labreze C, Lorette G, Mallet S, Martin L, Mazereeuw-Hautier J, Phan A, Plantin P, Quere I, Vabres P, Bourgoin H, Giraudeau B, Maruani A; Groupe de Recherche de la Societe Francaise de Dermatologie Pediatrique. Topical sirolimus 0.1% for treating cutaneous microcystic lymphatic malformations in children and adults (TOPICAL): protocol for a multicenter phase 2, within-person, randomized, double-blind, vehicle-controlled clinical trial. Trials. 2019 Dec 17;20(1):739. doi: 10.1186/s13063-019-3767-8. PMID 31847908